CLINICAL TRIAL: NCT05781178
Title: Analysis of the Aetiological Factors of Malnutrition: Inflammation and Oral Intake
Brief Title: Analysis of the Aetiological Factors of Malnutrition
Acronym: AFEDIN
Status: Completed | Type: Observational
Sponsor: Endocrinology and Clinical Nutrition Research Center, Spain (Other)
Collaborators: Adventia Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: PI23 3024
Record Dates: First submitted 2023-02-28; First posted 2023-03-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Disease-related Malnutrition; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Docosahexaenoic Acids; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement rich in omega-3 and olive oil polyphenols — Nutritional intervention with an oral nutrition supplement with anti-inflammatory effect and a programme of physical exercise
  Other Names: Physical activity

SUMMARY:
Disease-related malnutrition (DRM) is a frequent syndrome in clinical practice, in which the mutual relationship between disease and malnutrition is observed. Inflammation, anorexia, changes in body composition or in energy and protein requirements, contribute to the development of DRM. The Global Leadership Initiative on Malnutrition (GLIM criteria) provides a diagnostic system of malnutrition that has been accepted by the main international scientific societies in the field of clinical nutrition.

The GLIM criteria proposes an algorithm that includes phenotypic criteria (weight loss, underweight and low muscle mass), with their corresponding severity thresholds, and aetiological criteria (decreased oral intake, nutrient malabsorption and the presence of an inflammatory component). The diagnosis of malnutrition is established when an aetiological and a phenotypic criterion are met.

The aim of the study is to determine the diagnostic and prognostic value of aetiological factors of malnutrition based on GLIM criteria, presence and degree of inflammation and dietary intake, in patients diagnosed with DRM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DRM based on GLIM criteria with the presence of the aetiological criterion of inflammatory component and candidate for medical nutritional treatment according to current regulations.
* Agreeing to voluntarily participate in the study and sign the informed consent form, after having read the participant information sheet.
* Presence of an inflammatory response (CRP>3 mg/dl)
* Having an adequate cultural level and understanding of the clinical study.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with advanced liver cirrhosis or chronic hepatitis (Child=C scale)
* Patients with advanced neoplastic disease with life expectancy <6 months
* Patients with renal insufficiency with creatinine clearance less than 45 ml/min
* Severe infection in the last 3 weeks
* Taking antibiotic therapy at the time of inclusion, with the exception of prophylactic treatments
* Taking corticosteroids at the current time or one month prior to inclusion
* Treatment with biological therapies (antibodies) at the current time or one month in advance
* Taking non-steroidal anti-inflammatory drugs at the time of inclusion
* Taking omega 3 supplements for any concomitant pathology at the time of inclusion
* Undergoing surgery during the follow-up phase of the study
* Initiation of any drug during the study phase that may modify the patient's inflammatory pattern at the investigator's discretion
* Any criterion that, in the opinion of the principal investigator, could condition the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of DRM with the presence of an inflammatory response (CRP>3 mg/dl).
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Blood biochemistry data | Patients will be followed over a period of 3 consecutive months
  Albumin (g/dL)
Blood biochemistry data | Patients will be followed over a period of 3 consecutive months
  Prealbumin (mg/dL)
Blood biochemistry data | Patients will be followed over a period of 3 consecutive months
  C-reactive protein (mg/L)
Blood biochemistry data | Patients will be followed over a period of 3 consecutive months
  Ferritin (ng/mL)
Blood biochemistry data | Patients will be followed over a period of 3 consecutive months
  Neutrophils (x103/μL)
Blood biochemistry data | Patients will be followed over a period of 3 consecutive months
  Lymphocytes (x103/μL)
Blood biochemistry data | Patients will be followed over a period of 3 consecutive months
  Platelets (x103/μL)

SECONDARY OUTCOMES:
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  TBW (total body water, L)
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  ECW (extracellular water, L)
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  ICW (intracellular water, L)
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  FFM (lean mass, kg)
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  FM (fat mass, kg)
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  BCM (body cell mass, kg)
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  ASMM (appendicular skeletal muscle mass, kg)
Bioelectrical impedance data (model (50 kHz) | Patients will be followed over a period of 3 consecutive months
  SMI (skeletal muscle mass index, kg)
Functional parameters | Patients will be followed over a period of 3 consecutive months
  Test up and go (patient sits in a chair and is told to stand up (time starts), walks 3 meters, comes back and sits down (time ends). <20 seconds: OK; >20seconds: increased risk of falling
Functional parameters | Patients will be followed over a period of 3 consecutive months
  Dynamometry: hree measurements of the dominant hand will be made recording the mean and maximum, measured in kilograms. Jamar® dynamometers are most used in international studies and have several grip positions
Oral intake | Patients will be followed over a period of 3 consecutive months
  Energy: obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (kcal)
Oral intake | Patients will be followed over a period of 3 consecutive months
  Protein: obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (g)
Oral intake | Patients will be followed over a period of 3 consecutive months
  Carbohydrate: obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (g)
Oral intake | Patients will be followed over a period of 3 consecutive months
  Fat: obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (g)
Oral intake | Patients will be followed over a period of 3 consecutive months
  MUFA (monounsaturated fat acids): obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (g)
Oral intake | Patients will be followed over a period of 3 consecutive months
  PUFA (polyunsaturated fat acids): obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (g)
Oral intake | Patients will be followed over a period of 3 consecutive months
  EPA: obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (mg)
Oral intake | Patients will be followed over a period of 3 consecutive months
  DHA: obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (mg)
Oral intake | Patients will be followed over a period of 3 consecutive months
  Fibre: obtained from the nutritional analysis of a two-day dietary survey using the programme https://calcdieta.ienva.org (g)
Malnutrition Diagnosis | Patients will be followed over a period of 3 consecutive months
  GLIM criteria (Global Leadership Initiative on Malnutrition): GLIM rank indicates the patient's nutritional status according to 3 categories: well nourished, moderate malnutrition and severe malnutrition

CONTACTS AND LOCATIONS:
Overall Officials: Daniel de Luis Roman, Prof, Study Director — Endocrinology and Nutrition Department. Hospital Clínico Universitario de Valladolid (Spain); Samara Palma Milla, PhD, Principal Investigator — Endocrinology and Nutrition Department. Hospital Universitario La Paz (Spain); Alfonso Vidal Casariego, PhD, Principal Investigator — Endocrinology and Nutrition Department. Complejo Hospitalario Universitario de A Coruña (Spain); José M García Almeida, PhD, Principal Investigator — Endocrniology and Nutrition Department. Hospital Universitario Virgen de la Victoria (Spain)
Locations (15):
- Spain (15):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, A Coruña
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No